CLINICAL TRIAL: NCT05534750
Title: Evaluation of the Early Bactericidal Activity of Tedizolid and Linezolide Against Mycobacterium Tuberculosis
Brief Title: Evaluation of the Early Bactericidal Activity of Tedizolid and Linezolide Against Mycobacterium Tuberculosis (TEDITUB)
Acronym: TEDITUB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP210084
Record Dates: First submitted 2022-07-22; First posted 2022-09-09 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Tuberculosis; Multidrug Resistant Tuberculosis
Keywords: Tuberculosis; Multidrug Resistant; Linezolid; Tedizolid; Pyrazinamide; Rifampicin; Isionazid; Ethambutol; Early Bactericidal Activity
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — tedizolid phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tedizolid arm (Experimental): Patients will be taken 1 tablet per day of 200 mg film-coated of Tedizolid (SIVEXTRO®), in the morning for 7 days. Then, the early bactericidal activity will be measured and compared to the other arms.
  Interventions: Drug: Tedizolid arm (SIVEXTRO®)
- Linezolid arm (Experimental): Patients will be taken 2 tablets per day of 600 mg film-coated of Linezolid (ZYVOXID®) in the morning for 7 days. Then, the early bactericidal activity will be measured and compared to the other arms.
  Interventions: Drug: Linezolid arm (ZYVOXID®)
- Standard quadruple therapy arm (Active Comparator): Patients will be taken :
  ISONIAZIDE :
  o A dosage of 3 to 5mg / kg / day for 7 days (to be taken in the morning on an empty stomach) of Isoniazid (RIMIFON®)
  RIFAMPICINE :
  o A dosage of 10mg / kg / day for 7 days (to be taken in the morning on an empty stomach)
  ETHAMBUTOL :
  o A dosage of 15-20mg / kg / day for 7 days (to be taken in the morning on an empty stomach) of Ethambutol
  PYRAZAMIDE :
  o A dosage of 20-25mg / kg / day for 7 days (to be taken in the morning on an empty stomach) of Pyrazinamide
  Then, the early bactericidal activity will be measured and compared to the other arms.
  Interventions: Drug: Standard quadruple therapy arm

INTERVENTIONS:
Drug: Tedizolid arm (SIVEXTRO®) — Patients will be taken 1 tablet per day of 200 mg film-coated of Tedizolid (SIVEXTRO®), in the morning for 7 days. Then, the early bactericidal activity will be measured and compared to the other arms.
  Arms: Tedizolid arm
Drug: Linezolid arm (ZYVOXID®) — Patients will be taken 2 tablets per day of 600 mg film-coated of Linezolid (ZYVOXID®) in the morning for 7 days. Then, the early bactericidal activity will be measured and compared to the other arms.
  Arms: Linezolid arm
Drug: Standard quadruple therapy arm — Patients will be taken :
  ISONIAZIDE :
  o A dosage of 5mg / kg / day for 7 days (to be taken in the morning on an empty stomach) of Isoniazid (RIMIFON®)
  RIFAMPICINE :
  o A dosage of 10mg / kg / day for 7 days (to be taken in the morning on an empty stomach)
  ETHAMBUTOL :
  o A dosage of 15-20mg / kg / day for 7 days (to be taken in the morning on an empty stomach) of Ethambutol
  PYRAZAMIDE :
  o A dosage of 20-25mg / kg / day for 7 days (to be taken in the morning on an empty stomach) of Pyrazinamide
  Then, the early bactericidal activity will be measured and compared to the other arms.
  Arms: Standard quadruple therapy arm

SUMMARY:
The objective of this work is to measure the early bactericidal activity of tedizolid, to compare it with the bactericidal activity of linezolid (reference molecule for the treatment of multidrug-resistant tuberculosis) and with that of standard quadruple therapy (reference treatment of drug susceptible tuberculosis).

DETAILED DESCRIPTION:
This is a Phase 2, prospective, randomized, open-label controlled trial in 3 parallel groups comparing tedizolid with 2 standard treatments: linezolid (oxazolidinone whose anti-tuberculosis activity has already been demonstrated) and standard treatment for tuberculosis (quadruple therapy: isoniazid, rifampicin, ethambutol, pyrazinamide ). The objective is to measure the early bactericidal activity of tedizolid, to compare it with the bactericidal activity of linezolid and with that of standard quadruple therapy.

Design: A multicentric, open-label, randomized clinical trial

Sample size : 60 patients, 20 in each group

Treatments groups:

* Tedizolid arm:

  * Tedizolid (SIVEXTRO®),
  * 200 mg film-coated tablet
  * Dosage of 1 tablet per day to be taken in the morning for 7 days (taken with or without meals).
* Linezolid arm (ZYVOXID®):

  * Linezolid arm (ZYVOXID®)
  * 600 mg film-coated tablet
  * Dosage of 2 tablets per day to be taken in the morning for 7 days (taken with or without meals).
* Standard quadruple therapy arm:

  * Isoniazid (RIMIFON®) Tablets 50 or 200 mg Dosage 3 to 5mg / kg / day for 7 days to be taken in the morning on an empty stomach.
  * Rifampicin, dosage 10mg / kg / day for 7 days to be taken in the morning on an empty stomach.
  * Ethambutol 15-20mg / kg / day for 7 days to be taken in the morning on an empty stomach.
  * Pyrazinamide 20-25mg / kg / day for 7 days to be taken in the morning on an empty stomach.

Treatment duration : 7 days

Assessement:

After signing the consent, patients will be randomized, a sputum sample will be taken before the first drug intake. Then, patients will be treated for 7 days depending on the randomization group (tedizolid, linezolid or standard quadruple therapy). Daily, a sputum of at least 2 mL will be withdrawn from the patients for 7 days.

A consultation with blood test will be carried out on D30, date of the patient's end of participation.

No interim analysis is planned. Analysis will be performed at the end of the study after data review and freezing of database.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and <75 years old
* Woman on childbearing age should be on effective contraception during the duration of the study and up to 6 months after treatment; a mechanical contraception (use of condom) will be strongly recommended
* Male (effective contraception must be used during duration of the study and up to 3 months after treatment)
* Patient with a first infection with Mycobacterium tuberculosis of pulmonary localization suspected by the presence of a clinical pulmonary symptomatology, a chest X-ray or an abnormal chest computed tomography, and the positive microscopic examination of a sputum (AFB +, presence of AFB) with confirmation of tuberculosis by a genotypic test demonstrating no resistance to rifampicin, without clinical signs of extra-thoracic involvement
* State medical assistance application being processed ( If patient does not benefit from social security),
* Signature of informed consent

Exclusion Criteria:

* Resistance to one of the anti-tuberculosis drugs used detected by a genotypic test in accordance with the recommendations of the High Council of Public Health of 2015;
* History of anti-tuberculosis treatment (patients with a documented negative genotypic test for isoniazid and rifampicin resistance may be included)
* History of treatment in the previous two years with one of the antibiotics evaluated in this trial lasting more than one month;
* Absolute contraindication to the use of at least one of the test molecules (isoniazid, rifampicin, ethambutol, pyrazinamide, linezolid, tedizolid);
* Tuberculosis having, in the opinion of the investigator, severity criteria not allowing to wait 7 days before starting standard treatment (oxygenorequirement, severe immunosuppression, extra-pulmonary involvement, any sign of severity requiring treatment in intensive care unit);
* HIV-infected patient receiving protease inhibitors whose antiviral treatment cannot be changed and therefore cannot receive rifampicin; or any other drug contraindicated with one of the study treatments (the list of contraindicated drugs is detailed in the following non-inclusion criteria).
* Neoplastic pathology during treatment with chemo and / or radiotherapy;
* Decompensated cirrhosis;
* Pregnancy, desire to become pregnant, breast-feeding (for women of childbearing potential, contraception should be used for the duration of the study and up to 6 months after treatment, mechanical contraception will be strongly recommended and up to 3 months after treatment);
* Protected adults (under guardianship, curatorship) and under safeguard of justice
* Significant laboratory abnormalities (hemoglobin <9g / dl, polynuclear neutrophils <500 / mm3, platelets <50,000 / mm3, creatinine clearance <30ml / min, ASAT or ALAT> 3N, and total bilirubin> 3N)
* Hyperuricaemia
* Porphyria
* Optic neuritis or peripheral neuropathy
* BMI≤ 16 kg/m2
* Participation in other interventional research
* Current treatment with one or more medications contraindicated in combination with linezolid: Linezolid should not be used in patients treated with monoamine oxidase A or B inhibitors (for example: phenelzine, isocarboxacid, selegiline, moclobemide) or who received one of these products in the previous two weeks
* Current treatment with one or more medications contraindicated in combination with quadritherapy:
* Combination with bictegravir, cobicistat, daclatasvir, dasabuvir, delamanid, grazoprevir/elbasvir, protease inhibitors boosted by ritonavir, isavuconazole, ledipasvir, lurasidone, midostaurin, ombitasvir/paritaprevir, praziquantel, rilpivirine, sofosbuvir, velpatasvir, voriconazole, voxilaprevir
* Gastrointestinal topicals, antacids and adsorbents and salts and aluminum hydroxides

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the early bactericidal activity (EBA) of tedizolid (200mg / day) at the end of the first 2 days of treatment (D3). | Day 3
  The measurement will be done as follow: EABD1D3= (log10 number of CFU (CFU= colony forming unit) of M. tuberculosis on medium 7H11/mL of sputum on D1) - (log10number of CFU of M. tuberculosis on medium 7H11/mL of sputum on D3)/2.

SECONDARY OUTCOMES:
Evaluation of the early bactericidal activity (EBA) of tedizolid between Day 3 and Day 8 | Day 8
  The measurement will be done as follow: EBAD3D8= (log10 number of CFU (CFU=colony forming unit) of M. tuberculosis on medium 7H11/mL of sputum on D3) - ( log10 number of CFU of M. tuberculosis on medium 7H11/mL of sputum at D8)/5
Comparison of the early bactericidal activity (EBA) of tedizolid between Day 1 and Day 3 | Day 3
  Compare the early bactericidal activity of tedizolid 200 mg / day to that of linezolid 1200 mg / day between Day 1 and Day 3
Comparison of the early bactericidal activity (EBA) of tedizolid between Day 3 and Day 8 | Day 8
  Compare the early bactericidal activity of tedizolid 200 mg / day to that of linezolid 1200 mg / day between Day 1 and Day 3 and between Day 3 and Day 8
Comparison of the early bactericidal activity of tedizolid 200 mg / day to that of standard quadruple therapy between Day 1 and Day 3 | Day 3
  Compare the early bactericidal activity of tedizolid 200 mg / day to that of standard quadruple therapy between Day 1 and Day 3
Comparison of the early bactericidal activity of tedizolid 200 mg / day to that of standard quadruple therapy between Day 3 and Day 8 | Day 8
  Compare the early bactericidal activity of tedizolid 200 mg / day to that of standard quadruple therapy between Day 3 and Day 8
Tedizolid pharmacokinetics'measurement | 24hours
  To measure the total and free concentration of tedizolid measured at 0, 1, 3, 5 and 24hours
Evaluation of Tedizolid's tolerance on hemoglobin | 30 days
  Rate of patients with hemoglobin <9, g / dl, which will lead to premature discontinuation of the administration of the treatment
Evaluation of Tedizolid's tolerance on polynuclear neutrophils | 30 days
  Rate of patients with polynuclear neutrophils <500 / mm3, which will lead to premature discontinuation of the administration of the treatment
Evaluation of Tedizolid's tolerance on platelets | 30 days
  Rate of patients with platelets <30,000 / mm3 which will lead to premature discontinuation of the administration of the treatment
Evaluation of Tedizolid's tolerance on creatinine clearance | 30 days
  Rate of patients with creatinine clearance <30ml / min which will lead to premature discontinuation of the administration of the treatment
Evaluation of Tedizolid's tolerance on AST/ALT | 30 days
  Rate of patients with AST or ALT> 5N which will lead to premature discontinuation of the administration of the treatment
Evaluation of Tedizolid's tolerance on bilirubin | 30 days
  Rate of patients with total bilirubin> 5N which will lead to premature discontinuation of the administration of the treatment
Evaluation of Tedizolid's tolerance on dress syndrome | 30 days
  Rate of patients with dress syndrome which will lead to premature discontinuation of the administration of the treatment.
Evaluation of Tedizolid's tolerance on optic neuropathy | 30 days
  Rate of patients with optic neuropathy which will lead to premature discontinuation of the administration of the treatment
Evaluation of Tedizolid's tolerance on peripheral neuropathy | 30 days
  Rate of patients with rapidly progressive peripheral neuropathy, which will lead to premature discontinuation of the administration of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas VEZIRIS, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bacteriology department- Hôpital Saint-Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided